CLINICAL TRIAL: NCT06063343
Title: A First-in-human, Single-center, Placebo-controlled, Randomized, Double-blind Study in Healthy Subjects to Evaluate Safety, Tolerability, Pharmacokinetics, Food Effect and Interaction With Midazolam After Oral Single and Multiple Ascending Dosing of KAND145
Brief Title: Evaluation of Safety, Tolerability, Pharmacokinetics, Food Effect and Interaction With Midazolam in Healthy Volunteers After Oral Single and Multiple Ascending Dosing of KAND145
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novakand Pharma AB (Industry)
Collaborators: LINK Medical Research AB (Unknown); Q&Q Labs AB (Unknown); CRST Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KAN0008; 2023-503909-11-01 (Other: EUCT)
Record Dates: First submitted 2023-05-17; First posted 2023-10-02 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Part 1 - SAD: Up to 48 participants will be sequentially enrolled into up to 6 cohorts (8 participants per cohort). The first 2 participants in all cohorts will be randomized to KAND145 or placebo in a 1:1 ratio. The 6 remaining participants will be randomized to KAND145/placebo in a 5:1 ratio. FE-part: After a wash-out period of 6-14 days after dosing with KAND145/placebo, Cohort 1:3 will receive a second dose of KAND145/placebo (as per initial randomization) together with a meal.
  Part 2 - MAD: Up to 40 participants will be sequentially enrolled into up to 5 cohorts (8 participants per cohort). Participants in each cohort will be randomly assigned to KAND145 or placebo in a 3:1 ratio. Midazolam-part: Two cohorts will receive a single dose of 4 mg midazolam. After a wash-out period of 6-14 days, the participants will start dosing of KAND145/placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study and the allocation of treatments (KAND145 or placebo) will not be disclosed to the participants or to the personnel at the investigational site (except for an unblinded pharmacist), until the database has been locked.
  The KAND145 and placebo products will be delivered from the manufacturer to the investigational site in an unblinded fashion. At the site, the KAND145 and placebo products will be prepared for use by an unblinded pharmacist. The dosing syringes that will be handled by other site personnel will be blinded.
  The KAND145 oral solution is slightly yellowish and may have a bitter taste, while the matching placebo oral solution is colorless and tasteless. Therefore all dosing syringes will be amber-colored or masked to hide the appearance of the product, and participants will be asked to use a nose clamp during administration of KAND145/placebo.
  Treatment with midazolam (applicable for Cohort 2:1 and Cohort 2:2) will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KAND145 for SAD (Part 1) (Experimental): In Part 1, SAD of KAND145 will be administered to up to 6 cohorts. Six participants in each cohort will receive KAND145. The first cohort will receive a starting dose of 60 mg KAND145 which is expected to lead to an average drug plasma concentration (Cave) of 0.2 µM. The maximum dose will be chosen to achieve a Cave of 10 µM.
  Interventions: Drug: KAND145
- Placebo for SAD (Part 1) (Placebo Comparator): In Part 1, 2 participants per cohort in up to 6 cohorts will receive placebo at the same dosing frequency as detailed for the experimental arm.
  Interventions: Drug: Placebo
- KAND145 for MAD (Part 2) (Experimental): In Part 2, MAD of KAND145 will be administered to up to 5 cohorts. Six participants in each cohort will receive doses of KAND145 BID for 8 days. The first cohort will receive a dose of KAND145 which is expected to lead to a Cave of 2 µM. The maximum daily dose will be 3000 mg KAND145.
  Interventions: Drug: KAND145
- Placebo for MAD (Part 2) (Placebo Comparator): In Part 2, 2 participants per cohort in up to 5 cohorts will receive placebo at the same dosing frequency as detailed for the experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KAND145 — In Part 1 of the study, single ascending doses of KAND145 will be administered; in Part 2 of the study, multiple ascending doses (BID for 8 days) of KAND145 will be administered.
  Arms: KAND145 for MAD (Part 2); KAND145 for SAD (Part 1)
Drug: Placebo — Participants randomized to the placebo arms will receive placebo at the same dosing frequency as the experimental arms.
  Arms: Placebo for MAD (Part 2); Placebo for SAD (Part 1)

SUMMARY:
The goal of this study is to learn more about the study candidate drug, KAND145, when given to healthy volunteers. The study will consist of two parts. In Part 1, the goal is to find out if the study drug KAND145 is safe and tolerable after a single dose. First, a small group of participants will receive a liquid for swallowing containing a low dose of the study drug or a liquid for swallowing that does not contain any drug. If this is safe and tolerable, higher doses will be given to subsequent groups of participants. Additionally, the effect of food on the metabolism of the study drug will be studied. In Part 2, the goal is to find out how the body absorbs, distributes, and gets rid of the study drug when it is taken twice a day for 8 days. As in Part 1, first a liquid for swallowing containing a low dose of the study drug or a liquid for swallowing that does not contain any study drug will be given to a first group of participants; additional doses will then be given to subsequent groups of participants. Additionally, it will be studied if the study drug KAND145 affects the pharmacokinetics of the medicine midazolam.

DETAILED DESCRIPTION:
This is a Phase 1, first-in-human (FIH), single-center, placebo-controlled, randomized, double-blind study in healthy subjects to evaluate safety, tolerability, PK, food effect (FE) and interaction with midazolam after oral single ascending dosing (SAD; Part 1 of the study) and multiple ascending dosing (MAD; Part 2 of the study) of KAND145. A Safety Review Committee (SRC) will evaluate safety data from each dose cohort before proceeding with the subsequent cohort.

The study population will consist of healthy adult male and female volunteers. Up to 88 participants (up to 48 participants in Part 1, up to 40 participants in Part 2) are planned to be enrolled in the study, at one investigational site.

Part 1: In this part, participants receive single doses of KAND145 or placebo. Four ascending dose levels (cohorts) are planned; this may be extended with up to 2 optional dosing cohorts. In one cohort, a potential food interaction will be studied in the FE-part.

Part 2: In this part, participants receive KAND145 or placebo twice a day (BID) for 8 consecutive days. Two ascending dose levels (cohorts) are planned; this may be extended with up to 3 optional dose levels (cohorts). To find out whether KAND145 has an effect on CYP3A4-mediated drug metabolism, the interaction of KAND145/placebo with midazolam will be studied in two cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any other study specific procedures.
2. Body weight >50 kg.
3. BMI ≥19.0 and <30.0 kg/m^2 at screening.
4. Healthy male and female subjects aged >18 and <65 years at screening.
5. Male subjects must agree to use an adequate method of contraception; Male subjects who are heterosexually active must use a condom with their partner, from the time of IMP administration until 72 hours after dosing of IMP, AND from the time of IMP administration until 90 days after dosing of IMP at least one of the following highly effective contraception methods (as per the Clinical Trial Facilitation Group, guidelines, 21/09/2020 Version 1.1) must be used by their female sexual partner:

   1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal)
   2. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable)
   3. Intrauterine device
   4. Intrauterine hormone-releasing system
   5. Bilateral tubal occlusion or hysterectomy
   6. Vasectomized male Or if the male subject has a post-menopausal partner.
6. Female subjects must be of non-childbearing potential (defined as pre-menopausal females with a documented tubal ligation or hysterectomy or bilateral oophorectomy; or as post-menopausal females defined as 12 months' amenorrhea [in questionable cases, a blood sample with simultaneous follicle stimulating hormone 25-140 IU/L and estradiol <200 pmol/L is confirmatory]).

   Female subjects of childbearing potential may be included if it is their preferred and permanent lifestyle to abstain from heterosexual relationships, and if they agree to continue such abstinence and to avoid starting of a pregnancy during their study participation.
7. Willingness and ability to comply with study procedures, visit schedules, study restrictions and requirements.

Exclusion Criteria:

1. Present or known history of clinically significant cardio- or cerebrovascular, pulmonary, renal, hepatic, neurological, mental, metabolic, endocrine, hematologic, or gastrointestinal disorder, significant respiratory disease, sleep apnea, narcolepsy or any other major disorder that may interfere with the objectives of the study, as judged by the Investigator.
2. Any clinically significant abnormalities in physical examination, ECG (e.g., QTcF>450 ms for males/>460 ms for females), clinical chemistry, hematology, or urinalysis results at screening, as judged by the Investigator.
3. Clinically significant abnormal blood pressure, defined as systolic blood pressure above or equal to 160 mmHg and/or diastolic blood pressure above or equal to 90 mmHg at screening.
4. Pulse rate <45 beats per minute at screening.
5. Clinically significant illness within the 5 days prior to the administration of the IMP.
6. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody or human immunodeficiency virus.
7. Known or suspected current or history of (within the most recent 5 years) drug or alcohol abuse or positive screen for drugs of abuse test or positive alcohol breath test at screening visit or any time prior to randomization.
8. Smoking >5 cigarettes per day (or equivalent consumption of other nicotine-containing products), or inability to refrain from smoking or using other nicotine-containing products during the stay at the study clinic.
9. Subject who has received any investigational drug within the last 3 months before administration of IMP, or who has received any dose of KAND567 in a previous clinical study.
10. Plasma donation within 1 month of the screening visit, or any blood donation/blood loss >450 mL during the 3 months prior to the screening visit.
11. Use of the herbal remedy St. John's Wort during 2 weeks prior to administration of the IMP (induces cytochrome P450-3A4).
12. Use of prescribed medication during 2 weeks prior to the administration of the IMP (or longer if the prescribed medication has a half-life long enough to potentially expose the subject to any significant systemic exposure, as judged by the Investigator).
13. Use of over the counter drugs (including herbals) during 1 week prior to the administration of the IMP or need for concomitant medications during the study. However, use of the following may be allowed: occasional paracetamol for pain relief (up to 3 g per 24 hours), vitamin D (up to 20 μg per 24 hours), supplementation therapy with thyroxin, iron, calcium, folate, estrogen, vitamin B12, and other vitamins and minerals at recommended doses, as judged by the Investigator. Intake of preparations containing iron, calcium or other metal ions will not, however, be permitted in the 10 hours preceding and 4 hours following IMP intake. Thus, their use cannot be allowed during the treatment period of Part 2.
14. Female subjects: Positive pregnancy test at screening visit or at any time prior to dosing.
15. Investigator considers the subject unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Part 1: Safety - Adverse events | From dosing (Day 1) until last follow-up (10-14 days post-dosing)
  Frequency and severity of AEs will be determined.
Part 1: Safety - Vital signs | From dosing (Day 1) until last follow-up (10-14 days post-dosing)
  Measured by the occurrence of clinically abnormal vital signs. Unit of measure: percent change from baseline
Part 1: Safety - electrocardiogram (ECG) | From pre-dose (within 60 minutes) until 24 hours post-dose
  Measured by the occurrence of clinically abnormal ECG. Unit of measure: percent change from baseline
Part 1: Safety - Safety laboratory tests | From screening until last follow-up (10-14 days after dosing)
  Measured by the occurrence of clinically abnormal lab test results (routine clinical chemistry, haematology and urinalysis). Unit of measure: percent change from baseline.
Part 2: PK - Maximum plasma (peak) drug concentration (Cmax) | From pre-dose (within 60 minutes) until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) during steady state.
Part 2: PK - Time to reach Cmax following drug administration (tmax) | From pre-dose (within 60 minutes) until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) during steady state.
Part 2: PK - Area under plasma concentration-time curve AUCτ | From pre-dose (within 60 minutes) until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) during steady state
Part 2: PK - Average plasma drug concentration (Cave [AUCτ/12]) | From pre-dose (within 60 minutes) until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) during steady state
Part 2: PK - Terminal half-life (t½z) | From pre-dose (within 60 minutes) until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) during steady state.

SECONDARY OUTCOMES:
Part 1 - PK: Cmax | From Day 1 until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) after single doses.
Part 1 - PK: tmax | From Day 1 until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) after single doses.
Part 1 - PK: AUCinf | From Day 1 until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) after single doses.
Part 1 - PK: Cave (AUCinf/12 h) | From pre-dose (within 60 minutes) until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) after single doses.
Part 1 - PK: t1/2z | From Day 1 until 24 hours post-dose
  Assessed for KAND145 and KAND567(AM) after single doses.
Part 2 - Safety: AEs | From the day before the first dose (Day -1) until last follow-up (10-14 days after the last dose)
  Frequency and severity of AEs will be determined
Part 2 - Safety: Vital signs | From the day before the first dose (Day -1) until Day 8
  Measured by occurrence of clinically abnormal vital signs. Unit of measure: percent change from baseline
Part 2 - Safety: ECG | From Day -1 until Day 8
  Measured by the occurrence of clinically abnormal ECG. Unit of measure: percent change from baseline
Part 2: Safety - Safety laboratory tests | From Day -1 until last follow-up (10-14 days after the last dose)
  Measured by the occurrence of clinically abnormal lab test results (routine clinical chemistry, haematology and urinalysis). Unit of measure: percent change from baseline
Part 2 - PK: Cmax for midazolam | From Day 1 until Day 9 of the midazolam-part of the study
  Only applicable for participants in Cohort 2:1 and Cohort 2:2 that will participate in the midazolam-part of the study.
Part 2 - PK: tmax for midazolam | From Day 1 until Day 9 of the midazolam-part of the study
  Only applicable for participants in Cohort 2:1 and Cohort 2:2 that will participate in the midazolam-part of the study.
Part 2 - PK: AUCinf for midazolam | From Day 1 until Day 9 of the midazolam-part of the study
  Only applicable for participants in Cohort 2:1 and Cohort 2:2 that will participate in the midazolam-part of the study.
Part 2 - PK: t½z for midazolam | From Day 1 until Day 9 of the midazolam-part of the study
  Only applicable for participants in Cohort 2:1 and Cohort 2:2 that will participate in the midazolam-part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Schulz, Study Director — Novakand Pharma AB
Locations (1):
- Clinical Research Services Turku - CRST Oy, Turku, Finland